CLINICAL TRIAL: NCT05302427
Title: The Effect of Infant Massage on Infant Growth, Mother-Infant Attachment, and Maternal Self-Confidence
Brief Title: Infant Massage and Infant Growth, Mother-Infant Attachment, and Maternal Self-Confidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Zubeyde Ezgi Ercelik, Principal Investigator, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21-5.1t/53
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Growth; Attachment; Self-Confidence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage group (Experimental): The massage group will be shown live one-to-one baby massage training via Microsoft Teams by the researcher, and the mother will be asked to apply it to her baby at the same time. Baby massage training; It consists of leg massage, face-abdominal massage, arm-chest massage and back massage and will be completed in four weeks.
  Interventions: Behavioral: Infant Massage
- Control group (No Intervention): Infant massage training will not be given to the mothers of the babies in the control group until the 20th week.

INTERVENTIONS:
Behavioral: Infant Massage — The training will start with a leg massage in the first session and the mother will be asked to do this once a day until the next lesson. The next week, the new massage movement will be shown to the mother and the training will continue, and the mother will be told to do the application throughout the week by integrating it with the previous movement this time, and the four-week training will be completed in this way. After the training, which massage movement was taught to the mothers every week, the application pictures of this part will be sent and at the end of the four-week training, the baby massage video and the baby massage guide will be sent to the mothers by e-mail.
  Arms: Massage group

SUMMARY:
Touch is an essential element in the healthy growth and development of the baby. Infant massage is the best way to touch babies. In line with the literature review on the subject, it has been reported that infant massage supports growth and development in infants, improves attachment between mothers and babies and decreases the level of depression and anxiety in mothers.

With the coronavirus pandemic, quarantine decisions have been implemented all over the world. In addition to the stress brought on by their new roles, new mothers have to cope with the anxiety and stress of being a parent and babysitting during the pandemic period. During the pandemic process, it is seen that depression and anxiety levels increase in mothers who have given birth, and maternal attachment is negatively affected. Depression and anxiety in mothers negatively affect the cognitive, physical, social and emotional development of babies. It is very important to encourage practices that increase mother-infant interaction, such as infant massage, during the pandemic period.

The universe of the research will consist of mothers and their babies who were followed up in İzmir Karşıyaka No. 8 Gülay Kaymak Family Health Center and Karşıyaka No. 4 Bostanlı-2 Family Health Center between May 2021 and May 2022. The sample of the study is 38-42. It is planned to create babies born in the 4th week of pregnancy, with a birth weight of over 2500 grams and who have completed their fourth week (one month old) (n:60).

DETAILED DESCRIPTION:
The sense of touch is the most developed sense in newborns and is very important in perceiving the environment. The sense of touch in newborn babies is well developed throughout the body, especially on the tongue, lips, ears and forehead. When the baby is touched and held, he communicates with his environment and caregiver, and begins to recognize his environment. The sense of touch also positively affects the psychosocial development of babies. Infant massage is the best way to touch the baby. In recent years, research on infant massage has been the focus of the literature. When the literature is examined; it is seen that the positive effects of baby massage that support the growth and development of babies are proven by scientific research.

Attachment is defined as a situation that begins with the birth of the baby and has a predominant emotional aspect. The basic sense of trust formed between the mother and the baby in the early stages of life supports the psychosocial development of the baby. Touch, which is an effective method in providing and developing the interaction between the baby and the mother, affects the attachment positively. Infant massage is one of the easiest and most natural ways to develop mother-infant attachment. Studies show that infant massage strengthens the attachment between mothers and babies.

Baby massage also increases the mother's self-confidence in baby care. In the postpartum period, parents enter a new period in which they have to adapt to new roles, deal with baby care and the problems they experience with the baby. This period can sometimes cause problems such as lack of self-confidence, stress, anxiety and fear in mothers. The fear, anxiety and stress experienced by mothers regarding infant care can negatively affect mother-infant attachment. When the studies were examined, it was reported that the self-confidence score of the mothers who massaged was higher than the mothers in the control group in the study of with low birth weight babies and their mothers. In the qualitative study, mothers who apply baby massage defined massage as "a relaxing practice that provides emotional and physical contact with their babies". In addition, mothers stated that massage increased their self-confidence regarding the role of motherhood.

A newborn baby is born with about 100 billion neurons. Connections begin to form between neurons in the brain, especially in the first year after birth. While connections are formed with the warnings and experiences they receive throughout their lives; Neurons that do not receive enough stimulation die because they cannot make new connections. In babies who are given positive stimuli, intercellular connections are intense and their intelligence levels are positively affected. During the first two years of life, the rate of development of connections between neurons is quite high. Infant massage applied in these years contributes to the strengthening of the nervous system. The brain development of babies who are deprived of physical contact is adversely affected. Therefore, touch is an indispensable element in both the physical growth and development of the baby and the brain development.

In Turkey, no training is given on infant massage in family health centers. However, the positive effects of massage on babies and mothers have been demonstrated by scientific research. The role of nurses in mother-infant interaction is very important, making applications that support mother-infant interaction in the postpartum period and guiding mothers in this process is an important nursing practice. While nurses are training mothers, they should provide infant massage training within infant care routines, counsel mothers on infant massage and encourage them.

This study was designed in a randomized controlled, pre-test-post-test experimental model to examine the effects of infant massage on growth, mother-infant attachment, and mothers' self-confidence.

ELIGIBILITY:
Inclusion Criteria:

* The mother knows how to read, write and use a computer,
* The mother's consent to participate in the study,
* Babies 38-42. to be born at the gestational week and to have a birth weight of over 2500 grams and to have completed the fourth week.

Exclusion Criteria:

* Multiple pregnancy
* The mother has a disease or disability that prevents her from massaging her baby.

Ages: 4 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Maternal Attachment Inventory (MAI) | end of week 4
  The MAI is a 26-item self-report questionnaire used to measure mother-child attachment. Each item represents a maternal activity (e.g. 'I tell others about my baby') or feeling (e.g. 'I feel love for my child') which indicates affection towards the child. Items are scored on a 4-point Likert scale ranging from 1 (almost never)-4 (almost always). Total MAI scores range from 26-104, with higher scores indicating greater maternal attachment. The mean score of mother attachment inventory (pre-intervention assessment)
Maternal Attachment Inventory (MAI) | end of week 20
  The MAI is a 26-item self-report questionnaire used to measure mother-child attachment. Each item represents a maternal activity (e.g. 'I tell others about my baby') or feeling (e.g. 'I feel love for my child') which indicates affection towards the child. Items are scored on a 4-point Likert scale ranging from 1 (almost never)-4 (almost always). Total MAI scores range from 26-104, with higher scores indicating greater maternal attachment. The mean score of mother attachment inventory (post-intervention assessment)
Growth Parameter | end of week 4
  The mean of baseline weight (in grams)
Growth Parameter | end of week 8
  The mean change in body weight from end of week 4 to end of week 8 (in grams)
Growth Parameter | end of week 12
  The mean change in body weight from end of week 8 to end of week 12 (in grams)
Growth Parameter | end of week 16
  The mean change in body weight from end of week 12 to week end of 16 (in grams)
Growth Parameter | end of week 20
  The mean change in body weight from end of week 16 to week end of 20 (in grams)
Growth Parameter | end of week 4
  The mean of baseline body length (in centimeters)
Growth Parameter | end of week 8
  The mean change in body length from end of week 4 to end of week 8 (in centimeters)
Growth Parameter | end of week 12
  The mean change in body length from end of week 8 to end of week 12 (in centimeters)
Growth Parameter | end of week 16
  The mean change in body length from end of week 12 to end of week 16 (in centimeters)
Growth Parameter | end of week 20
  The mean change in body length from end of week 16 to end of week 20 (in centimeters)
Head circumference | end of week 4
  The mean of baseline head circumference (in centimeters)
Head circumference | end of week 8
  The mean change in head circumference from end of week 4 to end of week 8 (in centimeters)
Head circumference | end of week 12
  The mean change in head circumference from end of week 8 to end of week 12 (in centimeters)
Head circumference | end of week 16
  The mean change in head circumference from end of week 12 to end of week 16 (in centimeters)
Head circumference | end of week 20
  The mean change in head circumference from end of week 16 to end of week 20 (in centimeters)

SECONDARY OUTCOMES:
Pharis Self-Confidence | end of week 4
  The Pharis Self-Confidence Scale, which is a 13-item five-point measurement tool, measures a parent's feelings of self-confidence about daily baby care. Each infant care item is rated from 1 to 5 (not at all, very little, moderately, very much, completely). The increase in the total score obtained from the scale indicates that the self-confidence levels of the mothers increase in baby care. The lowest score on the "Pharis Self-Confidence" scale is 13, the highest score is 65.The mean score of pharis self-confidence (pre-intervention assessment)
Pharis Self-Confidence | end of week 20
  The Pharis Self-Confidence Scale, which is a 13-item five-point measurement tool, measures a parent's feelings of self-confidence about daily baby care. Each infant care item is rated from 1 to 5 (not at all, very little, moderately, very much, completely). The increase in the total score obtained from the scale indicates that the self-confidence levels of the mothers increase in baby care. The lowest score on the "Pharis Self-Confidence" scale is 13, the highest score is 65.The mean score of pharis self-confidence (pre-intervention assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Zübeyde Ezgi ERCELIK, MSc, Study Chair — Bandırma Onyedi Eylül University; Hatice BAL YILMAZ, Proffessor, Principal Investigator — Ege University
Locations (2):
- Turkey (Türkiye) (2):
  - Karşıyaka 4 No'lu Bostanlı- 2 Aile Sağlığı Merkezi, Izmir, Karşıyaka
  - Karşıyaka 8 Nolu Gülay Kaymak Aile Sağlığı Merkezi, Izmir, Karşıyaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vicente S, Verissimo M, Diniz E. Infant massage improves attitudes toward childbearing, maternal satisfaction and pleasure in parenting. Infant Behav Dev. 2017 Nov;49:114-119. doi: 10.1016/j.infbeh.2017.08.006. Epub 2017 Sep 1. PMID 28866286
- [Result] Gurol A, Polat S. The Effects of Baby Massage on Attachment between Mother and their Infants. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Mar;6(1):35-41. doi: 10.1016/j.anr.2012.02.006. Epub 2012 Mar 10. PMID 25030689
- [Result] Lu LC, Lan SH, Hsieh YP, Lin LY, Chen JC, Lan SJ. Massage therapy for weight gain in preterm neonates: A systematic review and meta-analysis of randomized controlled trials. Complement Ther Clin Pract. 2020 May;39:101168. doi: 10.1016/j.ctcp.2020.101168. Epub 2020 Apr 1. PMID 32379694
- [Derived] Ercelik ZE, Yilmaz HB. Effectiveness of infant massage on babies growth, mother-baby attachment and mothers' self-confidence: A randomized controlled trial. Infant Behav Dev. 2023 Nov;73:101897. doi: 10.1016/j.infbeh.2023.101897. Epub 2023 Nov 6. PMID 37939520
- See also: growth parameters — https://medicopublication.com/index.php/ijphrd/article/view/1415